CLINICAL TRIAL: NCT02591862
Title: Coversin in Paroxysmal Nocturnal Haemoglobinuria (PNH) in Patients With Resistance to Eculizumab Due to Complement C5 Polymorphisms
Brief Title: Coversin in Paroxysmal Nocturnal Haemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AKARI Therapeutics (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK578
Record Dates: First submitted 2015-09-10; First posted 2015-10-30 (Estimated); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2017-02

CONDITIONS: Paroxysmal Nocturnal Haemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — rEV576 protein, tick

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coversin (Nomacopan) (Other): This is an open label, non-comparator study.
  Patient will be given a single ablating dose of 0.57mg/kg per subject followed by daily repeat maintenance doses. The initial repeat dose will be 25% of the ablating dose. If this is insufficient to maintain complement inhibition at ≤10% of baseline (pre-treatment) level after 5 days of treatment the daily dose will be increased by doubling until that level of inhibition is achieved. In the event of 100% inhibition being achieved the dose may be titrated downwards at the PI's discretion until a satisfactory clinical result is obtained. If at any point in treatment complement inhibition falls to less than 50% of baseline a further ablating dose of 0.57mg/kg should be given. Coversin lyophilised powder in each vial was diluted with 0.6 mL water for injection prior to use.
  Interventions: Drug: Coversin

INTERVENTIONS:
Drug: Coversin — Patients enrolled in this protocol will initially be treated with an ablating dose of Coversin and daily repeat maintenance doses calculated according to body weight, the ablating dose to be 0.57mg/kg. Thereafter the daily repeat dose will be titrated according to clinical response and complement inhibition determined by CH50 ELISA. The initial repeat dose will be 25% of the ablating dose and this will be adjusted up or down if necessary once steady state is reached (5 days).
  Other Names: rVA576; rEV576

SUMMARY:
Coversin in Paroxysmal Nocturnal Haemoglobinuria (PNH) in patients with resistance to Eculizumab due to complement C5 polymorphisms.

DETAILED DESCRIPTION:
Coversin, a small protein complement C5 inhibitor which prevents the cleavage of C5 by C5 convertase into C5a and C5b, will be used in an open label, non-comparative clinical trial in patients with PNH and proven resistance to eculizumab due to C5 polymorphisms. Patients will be treated with Coversin by daily subcutaneous injection for 6 months in order to determine the safety and efficacy of the drug in these circumstances. If satisfactory control of the PNH is achieved, and at the discretion of the Principal Investigator (PI), patients will have the option of remaining on Coversin and being entered into the long term follow-up study for 2 years.

Please note, 'Coversin' is used throughout, but Nomacopan is the official name/INN.

Please note, the end points were assessed for 6 months, but the adverse events were measured over the 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Paroxysmal Nocturnal Haemoglobinuria (PNH)
* LDH >=1.5 Upper Limit of Normal (ULN)
* Resistance to Eculizumab proven by both a recognised C5 polymorphism on genetic screening and complement inhibition on CH50 ELISA of <100% at concentrations of Eculizumab in excess of 50 μg/mL
* Willing to self-inject Coversin daily or to receive daily subcutaneous injections by a home nurse or in a doctor's office or hospital clinic
* Males or females taking adequate contraceptive precautions if of childbearing potential, 18 - 80 years of age
* Body weight ≥50kg and ≤ 100kg
* The patient has provided written informed consent.
* Willing to avoid prohibited medications for duration of study
* Must agree to take appropriate prophylactic precautions against Neisseria infection.
* Must be counselled regarding the possible reproductive risks of using Coversin and be advised to use an adequate method of contraception pending further data on reproductive toxicology.

Exclusion Criteria:

* Body weight <50kg or>100kg
* Pregnancy (females)
* Failure to satisfy the PI of fitness to participate for any other reason
* Known allergy to ticks or severe reaction to arthropod venom (e.g., bee or wasp venom)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Dr Muus, Principal Investigator — Radboud University Medical Center; Saskia Dr Langemeijer, Study Director — Radboud University Medical Center
Locations (1):
- Dr Saskia Langemeijer, Nijmegen, Netherlands

REFERENCES:
- [Result] Schols S, Nunn MA, Mackie I, Weston-Davies W, Nishimura JI, Kanakura Y, Blijlevens N, Muus P, Langemeijer S. Successful treatment of a PNH patient non-responsive to eculizumab with the novel complement C5 inhibitor coversin (nomacopan). Br J Haematol. 2020 Jan;188(2):334-337. doi: 10.1111/bjh.16305. Epub 2019 Dec 16. No abstract available. PMID 31840801
- See also: Successful treatment of a PNH patient non-responsive to eculizumab with the novel complement C5 inhibitor coversin (nomacopan) — https://pubmed.ncbi.nlm.nih.gov/31840801/

RESULTS

PARTICIPANT FLOW:
Groups:
- Coversin: This is an open label, non-comparator study.
  Patient will be given a single ablating dose of 0.57mg/kg per subject followed by daily repeat maintenance doses. The initial repeat dose will be 25% of the ablating dose. If this is insufficient to maintain complement inhibition at ≤10% of baseline (pre-treatment) level after 5 days of treatment the daily dose will be increased by doubling until that level of inhibition is achieved. In the event of 100% inhibition being achieved the dose may be titrated downwards at the PI's discretion until a satisfactory clinical result is obtained. If at any point in treatment complement inhibition falls to less than 50% of baseline a further ablating dose of 0.57mg/kg should be given.
  Coversin: Patients enrolled in this protocol will initially be treated with an ablating dose of Coversin and daily repeat maintenance doses calculated according to body weight, the ablating dose to be 0.57mg/kg. Thereafter the daily repeat dose will be titrated according to clinical response and complement inhibition determined by CH50 ELISA. The initial repeat dose will be 25% of the ablating dose and this will be adjusted up or down if necessary once steady state is reached (5 days).
Period: Overall Study
Arm/Group | Coversin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Coversin
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 1
Weight [Number; unit: kg] | 67.8
Height [Number; unit: cm] | 172
Serum Lactate Dehydrogenase [Number; unit: U/L] | 1391
Haemoglobin concentration (Hb) [Number; unit: Millimole(s)/litre] | 8.2
Haptoglobin (Hp) concentration [Number; unit: Gram(s)/litre] | 0.0
Dependency on blood transfusion [Number; unit: participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Ratio of LDH to the Upper Limit of Normal (ULN)
Description: LDH is an indicator of disease progression in patients with PNH and is expected to fall to within 2x upper limit of normal (ULN) within 28 days in successfully treated patients. Units are measured in ratio of LDH:ULN, where the ULN is 250 U/L. The primary efficacy endpoint was the LDH AUC from Day 0 to 28 compared with 28 days pretreatment. Data for the 28 days pre-treatment was not collected, and as only one patient was recruited, the LDH values compared with baseline and the ratio of LDH to the Upper Limit of Normal (ULN) are presented.
Time Frame: Day 0 and Day 28
Population: Single arm trial design, results from 1 enrolled participant.
Measure: Number; unit: Ratio of LDH:ULN (250 U/L)
Groups:
- Coversin: This is an open label, non-comparator study.
  Patient will be given a single ablating dose of 0.57mg/kg per subject followed by daily repeat maintenance doses. The initial repeat dose will be 25% of the ablating dose. If this is insufficient to maintain complement inhibition at ≤10% of baseline (pre-treatment) level after 5 days of treatment the daily dose will be increased by doubling until that level of inhibition is achieved. In the event of 100% inhibition being achieved the dose may be titrated downwards at the PI's discretion until a satisfactory clinical result is obtained. If at any point in treatment complement inhibition falls to less than 50% of baseline a further ablating dose of 0.57mg/kg should be given.
  Coversin : Patients enrolled in this protocol will initially be treated with an ablating dose of Coversin and daily repeat maintenance doses calculated according to body weight, the ablating dose to be 0.57mg/kg. Thereafter the daily repeat dose will be titrated according to clinical response and complement inhibition determined by CH50 ELISA. The initial repeat dose will be 25% of the ablating dose and this will be adjusted up or down if necessary once steady state is reached (5 days).
Arm/Group | Coversin
Number analyzed (Participants) | 1
Ratio of LDH:ULN (250 U/L)
  Day 0 | 5.6
  Day 28 | 1.9

2. Primary Outcome: Number and Type of Adverse Events (AE)
Description: The number and type of reported AEs will be recorded as well as the opinion of the Principle Investigator (PI) as to their possible relationship to the study drug.
Time Frame: 2 years
Population: Results from 1 enrolled participant.
Measure: Number; unit: Events
Arm/Group | Coversin
Number analyzed (Participants) | 1
Events
  Serious Adverse Events (SAE) | 2
  Adverse Event (AE) (total) | 20
  Treatment Emergent Adverse Event (TAEA) | 13
  AE - moderate | 1
  AE - severe | 1
  AE- mild | 18

3. Secondary Outcome: Measurement of Haemoglobin (Hb) at Days 28, 90, and 180, Absolute and Change From Baseline
Description: Measuring change in mean Hb from Day 28, Day 90 and Day 180 (absolute and change from baseline)
Time Frame: Baseline, Day 28, Day 90 and Day 180
Population: Results from 1 enrolled participant.
Measure: Number; unit: millimole(s)/litre
Arm/Group | Coversin
Number analyzed (Participants) | 1
millimole(s)/litre
  Baseline | 8.2
  Day 28 (absolute) | 7.8
  Day 28 (change from baseline) | -0.7
  Day 90 (absolute) | 7.8
  Day 90 (change from baseline) | -0.4
  Day 180 (absolute) | 8.0
  Day 180 (change from baseline) | -0.2

4. Secondary Outcome: Measurement of Haptoglobin (Hp) at Days 28, 90 and 180, Absolute and Change From Baseline
Description: Measuring change in mean Hp from Day 28, Day 90 and Day 180 (absolute and change from baseline)
Time Frame: Baseline, Day 28, Day 90 and Day 180
Population: Results from 1 enrolled participant.
Measure: Number; unit: gram(s)/litre
Arm/Group | Coversin
Number analyzed (Participants) | 1
gram(s)/litre
  Baseline | NA — Haptoglobin was undetectable
  Day 28 | NA — Haptoglobin was undetectable
  Day 90 | NA — Haptoglobin was undetectable
  Day 180 | NA — The assay failed on day 180

5. Secondary Outcome: Measurement of Lactate Dehydrogenase (LDH) at Baseline, Day 90 and Day 180
Description: Measuring the change in LDH at Baseline, Day 90 and Day 180. LDH is an indicator of disease progression in patients with PNH and is expected to fall to within 2x upper limit of normal (ULN) within 28 days in successfully treated patients. Units are measured in ratio of LDH:ULN, where the ULN is 250 U/L.
Time Frame: Baseline, Day 90 and Day 180
Population: Single arm trial design, results from 1 enrolled participant.
Measure: Number; unit: Ratio of LDH:ULN (250 U/L)
Arm/Group | Coversin
Number analyzed (Participants) | 1
Ratio of LDH:ULN (250 U/L)
  Day 0 | 5.6
  Day 90 | 1.6
  Day 180 | 1.5

6. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy (FACIT) Score at Days 0, 28, 90 and 180
Description: Functional Assessment of Chronic Illness Therapy - fatigue (FACIT-F) is a 13 item instrument designed to assess fatigue/tiredness and it's impact on daily activities and functioning in a chronic disease setting. The scale for each question in relation to quality of life ranges from 0-4 where 0= not at all, 1= a little bit, 2= somewhat, 3 = quite a bit and 4= very much. An increase in the scale score indicates an improvement in quality of life (less fatigue). A maximum score of 52 is interpreted as no fatigue . Baseline is assumed as 0.0 to demonstrate the change in units.
  The subscale score (as presented) is determined as per FACIT-f guidance, by multiplying the sum of the item scores by the number of items in the subscale, then divide by the number of items answered.
Time Frame: Day 28, 90 and 180
Measure: Number; unit: FACIT-f scale (Change from Baseline)
Groups:
- Coversin: This is an open label, non-comparator study.
  Patient will be given a single ablating dose of 0.57mg/kg per subject followed by daily repeat maintenance doses. The initial repeat dose will be 25% of the ablating dose. If this is insufficient to maintain complement inhibition at ≤10% of baseline (pre-treatment) level after 5 days of treatment the daily dose will be increased by doubling until that level of inhibition is achieved. In the event of 100% inhibition being achieved the dose may be titrated downwards at the PI's discretion until a satisfactory clinical result is obtained. If at any point in treatment complement inhibition falls to less than 50% of baseline a further ablating dose of 0.57mg/kg should be given. Coversin lyophilised powder in each vial was diluted with 0.6 mL water for injection prior to use.
  Coversin: Patients enrolled in this protocol will initially be treated with an ablating dose of Coversin and daily repeat maintenance doses calculated according to body weight, the ablating dose to be 0.57mg/kg. Thereafter the daily repeat dose will be titrated according to clinical response and complement inhibition determined by CH50 ELISA. The initial repeat dose will be 25% of the ablating dose and this will be adjusted up or down if necessary once steady state is reached (5 days).
Arm/Group | Coversin
Number analyzed (Participants) | 1
FACIT-f scale (Change from Baseline)
  Day 28 | 13.0
  Day 90 | 13.3
  Day 180 | 11.0

7. Secondary Outcome: Change in Quality Of Life Questionnaire (QOQ) Score at Days 0, 28, 90 and 180
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 instrument measures the change in the quality of of life of patients in the trial. It comprises 30 questions on daily QOL and incorporates a global health status, five functional scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, nausea/vomiting, pain), and six single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). All of the scales range in score from 0 to 100, A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. Scale scores were calculated by averaging items within scales and transforming average scores linearly.
Time Frame: Day 28, 90 and 180
Population: Single arm trial design, results from 1 enrolled participant.
Measure: Number; unit: Scores on a scale (Change from baseline)
Arm/Group | Coversin
Number analyzed (Participants) | 1
Scores on a scale (Change from baseline)
  Global Health Status/ QOL (day 28) | 16.7
  Global Health Status/ QOL (day 90) | 16.7
  Global Health Status/ QOL (day 180) | 16.7
  Physical Functioning (day 28) | 6.6
  Physical Functioning (day 90) | 0.0
  Physical Functioning (day 180) | 6.6
  Role functioning (day 28) | 33.4
  Role functioning (day 90) | 33.4
  Role functioning (day 180) | 16.7
  Emotional functioning (day 28) | 16.6
  Emotional functioning (day 90) | 8.3
  Emotional functioning (day 180) | 8.3
  Cognitive functioning (day 28) | 33.3
  Cognitive functioning (day 90) | 16.7
  Cognitive functioning (day 180) | 16.7
  Social functioning (day 28) | 0.0
  Social functioning (day 90) | 0.0
  Social functioning (day 180) | 0.0
  Fatigue symptom scale (day 28) | -11.1
  Fatigue symptom scale (day 90) | 0.0
  Fatigue symptom scale (day 180) | 0.0
  Nausea and vomiting symptom scale (day 28) | 0.0
  Nausea and vomiting symptom scale (day 90) | 0.0
  Nausea and vomiting symptom scale (day 180) | 0.0
  Pain symptom scale (day 28) | 0.0
  Pain symptom scale (day 90) | 16.7
  Pain symptom scale (day 180) | 0.0
  Symptom: Dyspnoea (day 28) | 0.0
  Symptom: Dyspnoea (day 90) | 0.0
  Symptom: Dyspnoea (day 180) | 0.0
  Symptom: Insomnia (day 28) | -33.3
  Symptom: Insomnia (day 90) | 0.0
  Symptom: Insomnia (day 180) | 0.0
  Symptom: Appetite loss (day 28) | 0.0
  Symptom: Appetite loss (day 90) | 0.0
  Symptom: Appetite loss (day 180) | 0.0
  Symptom: constipation (day 28) | 0.0
  Symptom: constipation (day 90) | 0.0
  Symptom: constipation (day 180) | 0.0
  Symptom: diarrhoea (day 28) | -33.3
  Symptom: diarrhoea (day 90) | -33.3
  Symptom: diarrhoea (day 180) | -33.3
  Symptom: financial difficulties (day 28) | 0.0
  Symptom: financial difficulties (day 90) | 0.0
  Symptom: financial difficulties (day 190) | 0.0

8. Secondary Outcome: Dependency on Blood Transfusion
Description: Number of participants depending on blood transfusion prior to starting the study compared to during the study.
Time Frame: Day 0 through to study completion (2 years)
Population: Results from 1 enrolled participant.
Measure: Number; unit: participants
Arm/Group | Coversin
Number analyzed (Participants) | 1
participants
  Transfusion dependent prior to starting trial | 0
  Transfusion dependent during trial | 0

ADVERSE EVENTS:
Time Frame: Duration of the study (2 years)
Arm/Group | Coversin
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coversin (N=1)
Breakthrough Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coversin (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (5)
Injection site Reaction (General disorders) | 1 (13)
Malaise (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (6)
Insomnia (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemoglobinurea (Renal and urinary disorders) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Cold fingers and toes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI of the clinical units has independent rights of publication but will agree to discuss any intended publications or presentations with the Sponsor and to allow the Sponsor reasonable time to make comments, file or add to patent applications or request changes to the manuscript

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT02591862/Prot_SAP_000.pdf